CLINICAL TRIAL: NCT05508620
Title: A Phase Ib Study to Evaluate the Safety and Efficacy of Sirolimus for Injection (Albumin-bound) in Patients With Malignant Solid Tumors With TSC1/2 Genetic Alterations
Brief Title: A Study of Sirolimus for Injection (Albumin-bound) in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB1901-003
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Malignant Solid Tumors
MeSH Terms: interventions — Sirolimus; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sirolimus for Injection (Albumin-bound) (Experimental): Treatment with Sirolimus for Injection (Albumin-bound) will continue until disease progression, unacceptable toxicity, or other discontinuation criteria, whichever occurs first.
  Interventions: Drug: Sirolimus for Injection (Albumin-bound)

INTERVENTIONS:
Drug: Sirolimus for Injection (Albumin-bound) — Intravenous infusion

SUMMARY:
This is an open-label, multi-center phase 1b study to evaluate the safety and efficacy of Sirolimus for injection (albumin-bound) in patients with malignant solid tumors with TSC1 or TSC2 genetic alterations.

DETAILED DESCRIPTION:
This study will be conducted in two stages.

Stage 1: To evaluate the safety, tolerability and pharmacokinetics of Sirolimus for injection (albumin-bound), and determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). The Rolling-six design will be used for dose escalation.

Stage 2: To assess the antitumor activities of Sirolimus for injection (albumin-bound) in patients with malignant solid tumors harboring genetic alterations in TSC1 or TSC2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of malignant solid tumors, with TSC1 or TSC2 genetic alterations, and have no standard treatment or have failed standard treatments.
* Patients must have archival tumor tissues or agreed to have a tumor biopsy (if not, the sponsor's consent is required for enrollment).
* At least 1 measurable lesion as defined by RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Life expectancy of ≥3 months.
* Adequate marrow and organ function.
* Fasting serum triglyceride must be <300 mg/dL or <3.42 mmol/L; fasting serum cholesterol must be<350 mg/dL or <9.07 mmol/L.
* Fasting blood glucose must be<6.1 mmol/L and HbA1c< 6.5% in dose escalation, in other stage must be < 7.8 mmol/L and be< 8% respectively.
* Women of child-bearing potential, or men whose partners are women of childbearing age must agree to use reliable contraceptive methods during the trial period and at least 6 months after the last administration; women of childbearing age must have a negative serum pregnancy test within 7 days prior to the first administration, should not be breast feeding.
* Patients should understand and willingness to sign a written informed consent form prior to study entry.

Exclusion Criteria:

* Prior treatment with an mTOR inhibitor.
* Anti-tumor treatment within 4 weeks prior to first dose of study treatment.
* Participation in another therapeutic clinical trial with 4 weeks before study treatment.
* Major surgery within 4 weeks prior to study treatment, or have not fully recovered from any previous procedure.
* Unresolved toxicity from prior anti-tumor therapy greater than Grade 1 as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
* Patients with primary brain tumors or PEComa.
* Active uncontrolled or symptomatic central nervous system metastasis (CNS) or meningeal metastasis.
* History of serious cardiovascular disease.
* History of serious lung disease, such as interstitial lung disease and/or pneumonitis, or pulmonary hypertension, or pre-existing severely impaired lung function.
* Hydrothorax, ascites or pleural effusion with clinical symptoms or required treatment.
* Patients with hepatocellular carcinoma (HCC): Child-Pugh class B or C; or HCC with ≥50% liver occupation; or has a history or current evidence of hepatic encephalopathy; portal vein invasion at the main portal branch (Vp4).
* Live vaccine (including live attenuated vaccine) within 30 days before signing the informed consent.
* Infection that required systemic anti-infective therapy within 2 weeks before enrollment.
* History of autoimmune disease or immunodeficiency disease.
* Active Hepatitis B or Hepatitis C.
* Use of strong inhibitors or inducers of CYP3A4 within 2 weeks prior to start of treatment initiation, or requiring concomitant treatment during the study.
* Other server disease that may increase the risk of patients, or interfere the compliance of study procedures, or other reasons which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | At the end of Cycle 1 (each cycle is 21 days)
Recommended phase 2 dose (RP2D) | Up to 2 years
Overall response rate (ORR) | Up to 2 years

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 2 years
Duration of Response (DOR) | Up to 2 years
Progression-free Survival (PFS) | Up to 2 years
Overall survival (OS) | Up to 2 years
Maximum Plasma Concentration (Cmax) | Up to18 weeks
Time to reach maximum plasma concentration (Tmax) | Up to18 weeks
Area Under the Curve (AUC) | Up to18 weeks

IPD SHARING:
Plan to Share IPD: No